CLINICAL TRIAL: NCT05000619
Title: Encouraging Overdue Healthcare Appointment Scheduling Among Patients With Chronic Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Amir Goren, Program Director, Behavioral Insights Team, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2021-0442
Record Dates: First submitted 2021-08-02; First posted 2021-08-11 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Health Promotion; Prevention; Risk Reduction Behavior
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Participants will not be informed specifically of their assignment to different arms throughout the study. Providers who conduct appointments will not be randomized to study arms or informed of patient assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Outreach Postcard (Experimental): This group receives a postcard with a stock image on the front and a message encouraging regular visits to manage health on the back.
  Interventions: Behavioral: Outreach mailer
- Humorous Postcard (Experimental): This group receives a postcard with with a cartoon image and a visit-related joke on the front and a humorous message on the back, with additional information about why visits are important, and what to expect at the appointment.
  Interventions: Behavioral: Outreach mailer; Behavioral: Humor/Salience; Behavioral: Information
- Physician Letter (Experimental): This group receives a personalized letter signed by a physician with information about why visits are important, and what to expect at the appointment.
  Interventions: Behavioral: Outreach mailer; Behavioral: Doctor's authority; Behavioral: Information
- No-contact Control (No Intervention): This group will not receive a study mailer during the trial.

INTERVENTIONS:
Behavioral: Outreach mailer — Postcard or letter
  Arms: Humorous Postcard; Outreach Postcard; Physician Letter
Behavioral: Humor/Salience — Funny cartoon
  Arms: Humorous Postcard
Behavioral: Doctor's authority — Letter from a doctor
  Arms: Physician Letter
Behavioral: Information — Information about benefits of the appointment
  Arms: Humorous Postcard; Physician Letter

SUMMARY:
The goal of this study is to determine the most effective messages for encouraging patients with chronic conditions, who have not seen their doctor in at least one year, to return to the clinic. Study participants will receive postcards or letters encouraging them to make an appointment. Researchers will assess whether messages increase appointment scheduling (and attendance).

DETAILED DESCRIPTION:
About 18,500 Geisinger patients, Geisinger Health Plan members, and Medicaid patients with chronic illness have not been seen in a clinic for at least one year, which is concerning because regular appointments are necessary for chronic disease management. Geisinger is therefore working to encourage those with chronic illness and overdue appointments to return to the clinic.

In the present study, patients will either receive a mailer (with a message encouraging them to schedule an appointment with their physician), or no mailer. The purpose of the study is to compare three different mailers to assess which is most effective at encouraging patients to schedule and attend an appointment. The three mailers include (1) a standard outreach postcard (emphasizing that we are "checking in" with the patient), and, informed by behavioral science research, (2) a postcard with a cartoon and humorous messages and (3) a letter signed by a physician. The study will compare the effectiveness of the three experimental mailer arms to each other and to a no-contact control arm.

ELIGIBILITY:
Inclusion Criteria:

* Geisinger patient, Geisinger Health Plan member or Medicaid patient
* Chronic illness
* No appointment for > 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21562 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
Patients - Appointment scheduling | 30 days
  Proportion of Geisinger patients who schedule an appointment

SECONDARY OUTCOMES:
Patients - Appointment scheduling - Comparing mailers | 30 days
  Proportion of Geisinger patients who schedule an appointment, comparing relative efficacy of the mailers
Patients - Attendance at scheduled appointments within 180 days of mailer | 180 days
  Proportion of appointments (from the primary outcome) that were attended. This outcome focuses on attendance at appointments that were scheduled within 30 days of the mailer drop date.
  It is possible to schedule an appointment months in advance, so the Time Frame needs to be long to capture attendance at any appointment scheduled within 30 days of the mailer. 180 days should be sufficient to capture all scheduled appointments.
Patients, Members & Medicaid - Attendance at any appointment | 30 days
  Attendance at any appointment within 30 days of drop date
Patients, Members & Medicaid - Attendance at any appointment | 90 days
  Attendance at any appointment within 90 days of drop date
Patients, Members & Medicaid - Attendance at any appointment | 180 days
  Attendance at any appointment within 180 days of drop date
Patients, Members & Medicaid - Timing of appointment | 30 days
  Number of days between the drop date and any appointment captured in Secondary Outcome 3
Patients, Members & Medicaid - Timing of appointment | 90 days
  Number of days between the drop date and any appointment captured in Secondary Outcome 4
Patients, Members & Medicaid - Timing of appointment | 180 days
  Number of days between the drop date and any appointment captured in Secondary Outcome 5

OTHER OUTCOMES:
Patients - Appointment scheduling - Comparing mailers | 14 days
  Proportion of Geisinger patients who schedule an appointment, comparing relative efficacy of the interventions. Note: this analysis will inform internal operations but will not be reported in publication.
Patients - Calls to scheduling line | 30 days
  Proportion of Geisinger patients who call the appointment scheduling line.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Goren, PhD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with no personally identifiable information will be made available to other researchers on the Open Science Framework for transparency.
Supporting Information: SAP, Analytic Code
Time Frame: The data will become available after publication of study results in a scientific journal and will be available as long as the Open Science Framework hosts the data.
Access Criteria: The data on the Open Science Framework will be open to anyone requesting that information.
URL: http://osf.io

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-08-02): https://cdn.clinicaltrials.gov/large-docs/19/NCT05000619/SAP_000.pdf